CLINICAL TRIAL: NCT05089006
Title: Health Economic Assessment of Robot-assisted Surgery Compared to Open Surgery for Partial Nephrectomy in the Context of Renal Tumor
Brief Title: Cost-effectivness of Robot-assisted Surgery Compared to Open Surgery for Partial Nephrectomy in Context of Renal Tumor
Acronym: écoREIN
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Jacques HUBERT, Professeur, Central Hospital, Nancy, France
Other Study IDs: écoREIN
Record Dates: First submitted 2021-10-08; First posted 2021-10-22 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Renal Tumor
Keywords: kidney cancer; robot-assisted surgery; cost-effectiveness
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- robot-assisted surgery group: Patients undergoing robot-assisted surgery for small renal tumor
  Interventions: Procedure: Partial nephrectomy with robot-assisted and open surgery
- open surgery group: Patients undergoing open surgery for small renal tumor
  Interventions: Procedure: Partial nephrectomy with robot-assisted and open surgery

INTERVENTIONS:
Procedure: Partial nephrectomy with robot-assisted and open surgery — Robot-assisted partial nephrectomy (RAPN) is considered as a feasible minimally invasive alternative to open partial nephrectomy (OPN) for the surgical treatment of renal tumors. The main advantages of this technique include a three-dimensional magnified view of the surgical field, enhanced dexterity, and greater precision in both dissection and reconstruction.

SUMMARY:
This study aim to analyze cost-effectiveness of robot-assisted surgery compared to open surgery for partial nephrectomy in the context of renal tumor. A total of 400 patients were recruited in two centers in France corresponding to Reims(n=200) and Nancy hospital center (n=200). Patients recruited in Reims are corresponding to open surgery strategy, while patients of Nancy center are corresponding to robot-assisted surgery.

Costs analyzed included cost of intervention, hospital stay and complications. Effectiveness measure is corresponding to the rate of patients without acute complication at one year.

DETAILED DESCRIPTION:
The main objective of this study is to analyze cost-effectiveness of robot-assisted surgery compared to open surgery in the context of partial nephrectomy for renal tumor. Many studies demonstrated a better post-operative outcome with robot-assisted surgery mainly in terms of lower rate of complications. Results in terms of oncologic outcomes were equivalent. However, no study in France has analyzed the economic incentives of implementing robot-assisted surgery in the context of partial nephrectomy. It is very likely that the higher cost of robot-assisted surgery could be offset by a lower cost of post-operatives complications. The secondary purpose of this study is to analyze difference between robot-assisted and open surgery procedures in terms of operative time, hospital stay duration and rate of minor complications.

The study is based on a retrospective cohort of 400 patients. Half of patients (N=200) were recruited in Nancy hospital center and are corresponding to the robot-assisted surgery procedure. The other half is corresponding to open surgery arm and where recruited in Reims hospital center.

Inclusion criteria refer concerns patients over 18 years that were operated for minor renal tumor in Nancy and Reims hospital center. Patients operated for total nephrectomy were excluded from the analysis.

Data collected refers to the cost and effectiveness of the two compared procedures. Cost data are issued from hospital records and included the cost of hospital stay, surgical intervention and potential complications. Data related to effectiveness are obtained from patients medical records.

Cost-effectiveness analysis will be conducted to estimate the cost per one averted case of post-operative complication at one year. This consists on calculating the incremental cost-effectiveness ratio (ICER). Sensitivity analysis will be also conducted in order to estimate de confidence interval for the ICER.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing partial nephrectomy surgery for renal tumor
* Patients that gave informed consent for participating to the study

Exclusion Criteria:

* Patients undergoing partial nephrectomy surgery for other indication
* Patients that refused participation to the study
* Patients with horseshoe kidney
* Patients undergoing total nephrectomy for renal tumor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years old that undergone partial nephrectomy in Nancy and Reims center for small renal tumor.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2008-01-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Incremental cost-effectiveness ratio estimating cost per one acute post-operative complication averted | one year
  post-operative complication represents a relevant indicator in the context of renal nephrectomy. We aim to estimate the cost associated with one complication averted

SECONDARY OUTCOMES:
Difference in hospital stay duration between robot-assisted and open surgery | one year
  hospital stay represent a relevent indicator measuring effectiveness of intervention

IPD SHARING:
Plan to Share IPD: No
no personal data will be shared

REFERENCES:
- [Derived] Baghli A, Achit H, Audige V, Larre S, Branchu B, Balkau B, Eschwege P, Hubert J, Mazeaud C. Cost-effectiveness of robotic-assisted surgery vs open surgery in the context of partial nephrectomy for small kidney tumors. J Robot Surg. 2023 Aug;17(4):1571-1578. doi: 10.1007/s11701-023-01552-8. Epub 2023 Mar 15. PMID 36918464